CLINICAL TRIAL: NCT00341055
Title: A Pilot Study to Evaluate the Hematologic Response Rate of PROCRIT� (Epoetin Alfa) at 80,000 Units Once Weekly in Anemic Cancer Patients Receiving Chemotherapy
Brief Title: A Study to Evaluate the Hematologic Response Rate (the Rate at Which the Hemoglobin Level Rises) of PROCRIT (Epoetin Alfa) Given at a Dose of 80,000 Units Once Weekly to Cancer Patients With Anemia Who Are Receiving Chemotherapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005110
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Anemia; Cancer; Chemotherapy
Keywords: Anemia; Hemoglobin; Chemotherapy; Epoetin alfa
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the hematologic response, safety, and clinical outcomes of PROCRIT administered once a week in anemic cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
When comparing the proposed study dose to current literature, the initial study dose of 80,000 Units administered once per week is equivalent to an individual dose of 1142 Units/kg body weight for a 70 kg patient. It is also common in clinical practice for anemic cancer patients to be treated with a dose of PROCRIT (Epoetin alfa) of 40,000 Units weekly. This study was an open-label, non-randomized pilot study of cancer patients with non-myeloid malignancies with a hemoglobin < = 11 g/dL planned to receive at least 12 weeks of chemotherapy. The objective of the study was to evaluate the hematologic response, safety, and clinical outcomes of PROCRIT (Epoetin alfa) at 80,000 Units given subcutaneously (under the skin) once weekly in anemic cancer patients receiving chemotherapy. If, at any time the hemoglobin was > 13 g/dL, PROCRIT (Epoetin alfa) therapy was held until the hemoglobin was <= 12 g/dL, then resumed at 60,000 Units once weekly. The dose was also reduced if the hemoglobin rose by > 1.3 g/dL in a 2 week period.

Additionally, the incidence of anti-erythropoietin antibodies at baseline and at end of study/early withdrawal in study patients who have received a minimum of two or more doses of PROCRIT (Epoetin alfa) over at least a one-month period was evaluated. Rarely, antibodies to erythropoietin may form in patients who have some types of diseases (e.g., autoimmune diseases, rheumatoid arthritis, anemia of chronic disease) or in response to exposure to erythropoietin products such as Epoetin alfa necessitating discontinuation of the erythropoietin agent and medical treatment that may include blood transfusions. Hemoglobin level, vital signs (blood pressure) and occurrence and severity of adverse events was assessed throughout the study. PROCRIT (Epoetin alfa) was given at a dose of 80,000 Units subcutaneously (under the skin) for 12 weeks. The PROCRIT (Epoetin alfa) dose was monitored throughout the study and the dose was withheld or reduced as necessary to maintain hemoglobin level and rate of hemoglobin rise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of any non-myeloid malignancy planned to have received at least 12 weeks of chemotherapy with hemoglobin <= 11 g/dL
* Life expectancy > 6 months with Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Both male and female patients with reproductive potential must have used an adequate contraceptive method (e.g., abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment. Female patients with reproductive potential had a negative serum pregnancy test within 7 days of the first dose of study drug.

Exclusion Criteria:

* Previous radiation therapy to > 25% bone marrow reserve or planned radiation during study duration
* Packed red blood cells (PRBC) transfusion within 28 days of study entry
* Anemia due to factors other than cancer/chemotherapy, i.e., iron, folate, Vitamin B12 deficiency, hemolysis or GI bleeding
* Previous treatment with Epoetin alfa or any investigational forms of erythropoietin (e.g., gene-activated erythropoietin, novel erythropoiesis stimulating protein) within the previous 3 months
* uncontrolled hypertension or history of thrombotic vascular events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-06; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was major response defined as the proportion of patients with >= 2 g/dL hemoglobin (Hb) increase from baseline or Hb >= 12 g/dL and independent of transfusion within 28 days.

SECONDARY OUTCOMES:
The secondary efficacy endpoint was minor response defined as the proportion of patients with >= 1 g/dL hemoglobin (Hb) increase from baseline (up to 1.9 g/dL increase) and incidence of transfusion and independent of transfusion within 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Pilot Study to Evaluate the Hematologic Response Rate of PROCRIT (Epoetin alfa) at 80,000 Units Once Weekly in Anemic Cancer Patients Receiving Chemotherapy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=634&filename=CR005110_CSR.pdf
- See also: |Waltzman RJ, Williams D, Braly P. A Pilot Study to Evaluate the Safety and Clinical Outcomes of Once-Weekly Epoetin Alfa 80,000 U in Anemic Patients With Cancer Receiving Chemotherapy. Supportive Cancer Therapy. 2005;3(1):47-53 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=634&filename=CR005110_SupportiveCancerTherapy.pdf